CLINICAL TRIAL: NCT03183362
Title: Comparison of Barbed and Conventional Sutures in Adhesion Formation Following Cesarean Section; a Randomized Controlled Study
Brief Title: Comparison of Barbed and Conventional Sutures in Adhesion Formation Following Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Barbed sutures adhesions
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cesarean Section
Keywords: Barbed sutures,Cesarean Section, adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barbed suture ( STRATAFIX™ ) (Experimental): Cesarean section incision is closed using barbed sutures
  Interventions: Device: Barbed suture ( STRATAFIX™ )
- Conventional suture (VICRYL™) (Active Comparator): Cesarean section incision is closed using conventional sutures
  Interventions: Device: Conventional suture (VICRYL™)

INTERVENTIONS:
Device: Barbed suture ( STRATAFIX™ ) — Cesarean section incision will be closed using a 24-cm × 24-cm 0 polydioxanone double-armed suture on a 26-mm half-circle reverse cutting needle( STRATAFIX™ Spiral PDO Knotless Tissue Control Device, Ethicon Inc , Somerville, NJ, USA ).Patients who will return for a repeat caesarean (elective or emergency) will be evaluated intraoperatively for the presence of adhesions between various pelvic structures.
  Arms: Barbed suture ( STRATAFIX™ )
Device: Conventional suture (VICRYL™) — Cesarean section incision will be closed using 1-0 polyglactin 910 suture(VICRYL™.; Ethicon Inc, Sommerville, NJ) .Patients who will return for a repeat caesarean (elective or emergency) will be evaluated intraoperatively for the presence of adhesions between various pelvic structures .
  Arms: Conventional suture (VICRYL™)

SUMMARY:
The aim of this randomized controlled trial is to determine whether the use of barbed sutures to close uterine incision at cesarean section is associated with more postoperative adhesions compared with conventional sutures or not.

DETAILED DESCRIPTION:
The aim of this randomized controlled trial is to determine whether the use of barbed sutures to close uterine incision at cesarean section is associated with an increase in the rate of postoperative adhesions compared with conventional sutures or not. Primigravida patients undergoing transverse lower segment cesarean section will be included in the study.Cesarean section incision will be closed with double layers of continuous barbed or conventional sutures.Patients who will return for a repeat caesarean (elective or emergency) will be evaluated intraoperatively for the presence of adhesions between various pelvic structures.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida patients undergoing transverse lower segment cesarean section

Exclusion Criteria:

* Previous laparotomies
* Postoperative fever
* Patients with preterm pregnancies or in labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Adhesions formation rate | Through study completion, an average of 3 year
  Patients who will return for a repeat caesarean (elective or emergency) will be evaluated intraoperatively for the presence of adhesions between various pelvic structures.

CONTACTS AND LOCATIONS:
Overall Officials: Usama M. Fouda, Prof., Study Chair — Cairo University; Mohamed Zayed, Prof., Study Chair — Cairo University
Locations (1):
- Faculty of medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No